CLINICAL TRIAL: NCT03517930
Title: A Randomized, Crossover Manufacturing Transfer Study Comparing the Bioequivalence of a Single Oral Dose of Claritin-D® 12-Hour Extended Release Tablet (Loratadine 5mg/Pseudoephedrine Sulfate 120 mg, Manufacturer-SAG) to a Single Oral Dose of Claritin-D® 12-Hour Extended Release Tablet (Loratadine 5 mg/Pseudoephedrine Sulfate 120 mg, Manufacturer-Heist) Under Fasted Conditions in Healthy Adult Subjects
Brief Title: A Manufacturing Transfer Study Comparing the Bioequivalence of a Single Oral Dose of Claritin-D 12-Hour Extended Release Tablet From 2 Different Manufacturers Under Fasted Conditions in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19625
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Clinical Pharmacology
Keywords: Upper respiratory allergy symptoms including congestion
MeSH Terms: interventions — Loratadine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test treatment (Experimental): Healthy adult subjects under fasted conditions
  Interventions: Drug: Loratadine + Pseudoephedrine sulfate (Claritin-D, BAY818725) (Manufacturer-SAG); Drug: Loratadine + Pseudoephedrine sulfate (Claritin-D, BAY818725) (Manufacturer-Heist)
- Reference treatment (Active Comparator): Healthy adult subjects under fasted conditions
  Interventions: Drug: Loratadine + Pseudoephedrine sulfate (Claritin-D, BAY818725) (Manufacturer-SAG); Drug: Loratadine + Pseudoephedrine sulfate (Claritin-D, BAY818725) (Manufacturer-Heist)

INTERVENTIONS:
Drug: Loratadine + Pseudoephedrine sulfate (Claritin-D, BAY818725) (Manufacturer-SAG) — Oral, Loratadine 5 mg/ pseudoephedrine sulfate 120 mg (x1)
Drug: Loratadine + Pseudoephedrine sulfate (Claritin-D, BAY818725) (Manufacturer-Heist) — Oral, Loratadine 5 mg/ pseudoephedrine sulfate 120 mg (x1)

SUMMARY:
To evaluate the bioequivalence of one extended release combination (loratadine 5 mg/pseudoephedrine sulfate 120 mg) tablet manufactured for Bayer HealthCare LLC by SAG Manufacturing, S.L.U. Madrid, Spain (test treatment) to the extended release combination (loratadine 5 mg/pseudoephedrine sulfate 120 mg) tablet manufactured for Bayer SA-NV by Schering-Plough Labo NV Heist (reference treatment) which is currently marketed in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women
* Age 18 to 55 years inclusive
* Body mass index 18.5 to 30.0 kg/m*2 inclusive

Exclusion Criteria:

* Positive alcohol or drug screen at Screening or on Day -1 of each dosing period;
* Use of within 1 month before first study drug administration, systemic or topical medicines or substances which might affect the study objectives, any drug known to induce cytochrome P3A4/5 or P Glycoprotein (e.g., rifampin, carbamazepine, St. John's wort); Any drug known to inhibit cytochrome P3A4/5 or P Glycoprotein (e.g., clarithromycin, chloramphenicol, ketoconazole);
* History of hypersensitivity symptoms with the use of loratadine, desloratadine (Clarinex), or pseudoephedrine;
* Females who are pregnant or lactating
* Known severe allergies (e.g., allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids);
* More than moderate alcohol consumption (>40 g of alcohol regularly per day);
* Any history or suspicion of barbiturate, amphetamine, benzodiazepine, cocaine, opiates, methamphetamine or cannabis abuse;
* Loss of blood of 50 mL to 499 mL within 30 days of the first dose of trial treatment, or in excess of 500 mL within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis or injury)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlast) of loratadine and pseudoephedrine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Area under the curve from time 0 to the last measurable concentration.
Cmax of loratadine and pseudoephedrine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Maximum observed plasma level

SECONDARY OUTCOMES:
CL/F for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Total body oral clearance
Number of participants with adverse event | Up to 26 days
%AUC(tlast-∞) for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Percentage of AUC from last data point > lower limit of quantification (LLOQ) to infinity
Tmax for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Time at which Cmax is observed
Tlast for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Time point for last measurable concentration.
λz for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Terminal elimination rate constant
t1/2 for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Half-life
AUC(0-tlast) for desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Area under the curve from time 0 to the last measurable concentration.
Cmax for desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Maximum observed plasma level
AUC for loratadine, pseudoephedrine and desloratadine | Baseline (within 60 minutes of dosing) and at 15, 30, 45, 60 minutes and 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose in each treatment period
  Area under the curve from time 0 to infinity.

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services, Secaucus, New Jersey, United States